CLINICAL TRIAL: NCT03832634
Title: Fetal Genome Profiling After Non-Invasive Isolation of Trophoblast Cells
Brief Title: Fetal Genome Profiling Via Trophoblast Cells
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of personnel and funding resources
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1703018076
Record Dates: First submitted 2019-01-09; First posted 2019-02-06 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fetal Genome Profiling (Other): Trophoblast cells will be collected from the cervix approximately 5-6 weeks once pregnancy is achieved.
  Interventions: Diagnostic Test: Fetal Genome Profiling.

INTERVENTIONS:
Diagnostic Test: Fetal Genome Profiling. — Once pregnancy is achieved, patients will undergo non-invasive collection of trophoblast cells (trophoblast retrieval and isolation from the cervix, TRIC) at an early gestational age, approximately 5-6 weeks. The patient will also be screened with blood work for carrier status for genetic conditions.

SUMMARY:
The objective of this study is to utilize trophoblast cells accumulating in the endocervical canal at the beginning of pregnancy for non-invasive prenatal testing. If we are able to validate that trophoblast cells obtained at an early gestational age can be reliably used for prenatal testing, there is great potential to improve early pregnancy management and counseling options for potential parents. The target population will be all women between the age of 18-45 undergoing care at the Center for Reproductive Medicine (CRM) in order to achieve a pregnancy.

DETAILED DESCRIPTION:
The primary purpose of the study is to validate trophoblast retrieval and isolation from the cervix (TRIC) as a means of reliable non invasive prenatal genetic diagnosis (for both chromosomal abnormalities, as well as single gene defects).

The study population will be recruited from women, age 18 to 45, presenting to the Center for Reproductive Medicine (CRM) for medical care with the desire to become pregnant. Patients that achieve pregnancy will be invited by a physician to participate in the study. If prospective subjects agree to participate, they will meet with a co-investigator to go through the informed consent process.

Subjects will undergo a one-time non-invasive collection of trophoblast cells (trophoblast retrieval and isolation from the cervix, TRIC) at approximately 5-6 weeks of pregnancy as the experimental procedure for the study. TRIC is performed with ThinPrep kits using a cytobrush, the same method of Pap smear collection which is a routine part of prenatal care. The fetal trophoblast cells will then be isolated using immunomagnetic isolation. Once isolated, DNA fragmentation, fluorescent in situ hybridization (FISH), and single-cell PCR methods will be utilized to analyze the fetal genome at single nucleotide resolution. Any abnormal results identified by TRIC will be communicated to the subjects' by their physician in the office who will counsel them on the potential meaning of the results and recommend follow up testing to be ordered by their obstetrician to confirm results.

The cellular analysis from TRIC will then be compared to results obtained from CVS, amniocentesis, preimplantation genetic screening (PGS) and/or preimplantation genetic diagnosis (PGD) of the transferred embryo(s), or cytogenetic testing of fetal tissue in the event of miscarriage or pregnancy termination for validation. In the event that a patient does not undergo any of the aforementioned testing, TRIC results will be compared to birth outcomes.

Subjects will be followed via medical records through the final outcome of the pregnancy, whether termination of pregnancy, miscarriage, or live birth. If the pregnancy results in termination of pregnancy or miscarriage, cytogenetic testing of the fetus will be completed as standard care with the results compared to those obtained through TRIC testing. If the pregnancy results in live birth, basic neonatal information will be obtained via medical records, specifically whether the neonate is diagnosed with a disorder that can be identified through single gene testing (see attached table).

ELIGIBILITY:
Inclusion Criteria:

* Women 18 to 45 who achieve a pregnancy during study time period.
* If pregnancy result in miscarriage, cytogenetic testing must be completed on the product of conception.

Exclusion Criteria:

* Women whose cervical sample collection containing inadequate number of trophoblast cells for analysis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 1 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-02-14 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of chromosomal anomalies as detected via fetal genome analysis of trophoblast cells | 6 weeks post pregnancy
  Trophoblast cells isolated from the cervix will be used to detect chromosomal anomalies occurrences as a means of non-invasive prenatal screening.

SECONDARY OUTCOMES:
Occurrence of chromosomal anomalies detected via trophoblast cell analysis as compared to occurrence of chromosomal anomalies detected via preimplantation genetic testing (PGT), chorionic villi sampling (CVS), amniocentesis, or cytogenetic results. | 16 weeks post pregnancy
  Occurrence of chromosomal anomalies detected via trophoblast cells analysis will be compared to the occurrence of chromosomal anomalies detected via either PGT, CVS, amniocentesis, or cytogenetic which ever is available for validation.

CONTACTS AND LOCATIONS:
Overall Officials: Kangpu Xu, PhD, DVM, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No